CLINICAL TRIAL: NCT01455376
Title: Effect of Exogenous Lactate Infusion on Neurocognitive Function of Patients With Mild Traumatic Brain Injury
Brief Title: Effect of Exogenous Lactate on Neurocognitive in Brain Trauma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Padjadjaran (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AN-001.2011
Record Dates: First submitted 2011-10-05; First posted 2011-10-19 (Estimated); Last update posted 2011-10-21 (Estimated); Status verified 2011-10

CONDITIONS: Traumatic Brain Injury
Keywords: brain injury; cognitive function; sodium lactate; MMSE score
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hyperosmolar sodium chloride (No Intervention): Patients in this group received intravenous infusion of hyperosmolar Sodium Chloride 3% at 1.5 ml.KgBW-1 within 15 minutes before neurosurgery
- Hyperosmolar sodium lactate (Experimental): Patients in this group received intravenous infusion of hyperosmolar sodium lactate at 1.5 ml.KgBW-1 within 15 minutes before neurosurgery
  Interventions: Drug: hyperosmolar sodium lactate

INTERVENTIONS:
Drug: hyperosmolar sodium lactate — Patients in this group received intravenous infusion of hyperosmolar sodium lactate at 1.5 ml.KgBW-1 within 15 minutes before neurosurgery
  Other Names: Totilac
  Arms: Hyperosmolar sodium lactate

SUMMARY:
Mild traumatic brain injury (TBI) is the most common type of brain injury. Post-mild TBI disability could stem from cognitive, physical, psychological and social dysfunction which resulted in significant disability and unemployment. Long-term behavioral impairments which affected the individual's occupation, lifestyle, and family frequently occurred in individuals with mild to moderate brain injuries who physically fully recovered. In-vitro and in-vivo studies showed a better recovery of cognitive function after administration of exogenous lactate in traumatic brain injury. Therefore, this study is aimed to evaluate the effect of exogenous lactate infusion contained in hyperosmolar sodium lactate solution on cognitive function assessed by Mini Mental State Examination(MMSE)scale.

DETAILED DESCRIPTION:
Mild traumatic brain injury (TBI) is the most common type of brain injury. Post-mild TBI disability could stem from cognitive, physical, psychological and social dysfunction which resulted in significant disability and unemployment. Cognitive impairment post traumatic brain injury is due to the disruption of brain vascular bed and microstructural damage. Currently, there is no specific therapy for individual with mild TBI. Neuropsychological assessment and early management immediately after mild traumatic brain injury have been shown to reduce long term cognitive disability. In-vitro and in-vivo studies showed a better recovery of cognitive function after administration of exogenous lactate in traumatic brain injury.

The role of lactate in cerebral energy metabolism has been investigated widely. The ability of lactate as the sole energy substrate to support synaptic function has been demonstrated by different studies. In many studies, lactate has been proven to be a preferred or even an obligatory substrate over glucose for aerobic energy production during the initial stage of recovery from cerebral ischemia or hypoxia for recovery from ATP-depleted synaptic function and exogenously supplied lactate can support the early recovery of synaptic function after hypoxia.

However, the clinical studies evaluated the effect of lactate administration on cognitive function in patients with mild traumatic brain injury are still limited. Therefore, we conduct a study to evaluate the effect of exogenous lactate infusion contained in hyperosmolar sodium lactate solution on cognitive function assessed by Mini Mental State Examination (MMSE) score evolution in mild traumatic brain injury compared with patients receiving hyperosmolar sodium chloride 3 % as a control group. MMSE score can be used as a tool to describe cognitive function.

ELIGIBILITY:
Inclusion Criteria:

* Mild traumatic brain injury
* Glasgow Coma Scale (GCS) of 14-15
* Requires emergency neurosurgery procedures
* Physical status ASA I-II
* Onset of trauma < 9 hours

Exclusion Criteria:

* Multiple injury
* Pregnancy/lactation
* History of alcohol or barbiturate consumption prior to the injury

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2010-03; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Changes in neurocognitive function | 24 hours, 30 days, and 90 days post surgery
  The investigators evaluate the changes in neurocognitive function at several time points (24 hours, 30 days, and 90 days post surgery) using Mini Mental State Examination (MMSE) score in both groups. Osmolality and sodium level are also recorded in order to confirm that hyperosmolar sodium lactate is safe for traumatic brain injury patients

CONTACTS AND LOCATIONS:
Overall Officials: Tatang Bisri, MD,PhD,Prof, Principal Investigator — Faculty of Medicine Universitas Padjadjaran - Dr. Hasan Sadikin Hospital Bandung
Locations (1):
- Hasan Sadikin Hospital, Bandung, West Java, Indonesia